CLINICAL TRIAL: NCT00151294
Title: A Double-Blind, Placebo-Controlled Investigation Into the Safety and Efficacy of Escitalopram for Depression in Multiple Sclerosis
Brief Title: The Efficacy and Safety of Escitalopram for Depression in Multiple Sclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LXP-MD 45; 0410007546
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Depression; Multiple Sclerosis
Keywords: Depression (mild to moderate); Affective symptoms; Emotional lability; Multiple Sclerosis
MeSH Terms: conditions — Depression; Multiple Sclerosis; Affective Symptoms

INTERVENTIONS:
Drug: escitalopram oxalate antidepressant

SUMMARY:
Emotionally labile, depressed participants with multiple sclerosis treated with escitalopram will have a greater reduction in emotional lability scores and in their psychological distress scores than those who are randomized to receive placebo.

DETAILED DESCRIPTION:
Patients with multiple sclerosis who are experiencing mood lability and symptoms of depression will be randomized to receive either escitalopram 10mg/day or placebo tablets for a period of 6 weeks. It is hypothesized that patients receiving medication will experience a greater normalization of their emotional instability and a greater reduction in their depressive symptoms at the end of the six-week trial than those who are not receiving medication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple sclerosis
* Having mild to moderate depressive symptoms, with or without emotional lability
* Experiencing psychological distress

Exclusion Criteria:

* Meeting DSM-IV diagnostic criteria for Major Depressive Disorder or another Axis 1 diagnosis
* Cognitive impairment
* The presence of an unstable medical illness that might preclude completion of the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-11; Study Completion 2006-10

PRIMARY OUTCOMES:
Escitalopram-treated MS patients will have greater reductions in their depressive symptom scores than patients randomized to placebo
Adverse events for both groups will be similar

SECONDARY OUTCOMES:
Escitalopram-treated emotionally labile patients with MS will have a greater reduction in emotional lability scores than those randomized to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Barnett S Meyers, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork Presbyterian Hospital, White Plains, New York, United States